CLINICAL TRIAL: NCT05635812
Title: Brain and Eye Markers of Facial Expression Recognition and Disorders Associated with Autistic Symptoms
Acronym: MARQUEURS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: PINOIT 2022
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Brain Markers
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Participants Autism Spectrum Disorders (ASD): ASD according to DSM-5 criteria
  Interventions: Other: Neuropsychological assessment; Other: EEG experimentation; Other: Oculometry experimentation
- Participants 22q11.2: Participants with a genetic syndrome diagnosed by FISH or CGH-array
  Interventions: Other: Neuropsychological assessment; Other: EEG experimentation; Other: Oculometry experimentation
- Neurotypical participants: Neurotypical development
  Interventions: Other: Neuropsychological assessment; Other: EEG experimentation; Other: Oculometry experimentation

INTERVENTIONS:
Other: Neuropsychological assessment — neuropsychological assessment and clinical scales duration: 3 hours
Other: EEG experimentation — duration: 1 hour
Other: Oculometry experimentation — duration: 30 minutes

SUMMARY:
In everyday life, it is necessary to adjust one's behavior and reactions in order to interact and communicate with others in an appropriate manner. This adaptation is done by taking into account the emotions of the people with whom we interact. This reading of emotions is done by using visible clues on the face, in particular by observing the eye area of the interlocutor.

The aim of the study is to investigate how processes such as attention or memory influence emotion recognition, as well as (i) their alteration in the disease, and (ii) their link with the emergence of autistic and/or psychotic symptoms. We also want to study the implementation of compensatory strategies (used to compensate for difficulties in recognizing or perceiving emotions) and the link between the correct use of these strategies and the emergence of autistic and/or psychotic symptoms.

The present project plans to include a total of 120 participants: 30 participants with ASD, 30 patients with a particular genetic deletion 22q11.2 and 60 control participants.

After the inclusion visit, participation in the study will be divided into two half-days in order to perform a neuropsychological assessment, an EEG study and an oculometry study.

ELIGIBILITY:
Inclusion Criteria:

* Person, and if necessary his or her legal representative, who has given his or her non-objection
* Person whose mother tongue is French.
* Person aged between 7 and 50 years old.
* Person diagnosed with ASD according to DSM-5 criteria, person with a genetic syndrome diagnosed by FISH or CGH array (22q11 deletion), person with typical development matched in age and gender.
* Psychotropic treatment unchanged for one month and stable symptomatology.

Exclusion Criteria:

* Recent addiction according to DSM-5 criteria, excluding tobacco.
* Pregnant women.
* Uncorrected visual acuity disorder.
* Use of somatic or psychic medication that may alter brain/psychic functioning (e.g. corticosteroids).
* Neurological disorder of vascular/infectious or neurodegenerative origin.

Ages: 7 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: ASD, 22q11.2 and neurotypical participants
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Electrical brain activity in response to visual stimulation measured by electroencephalography | at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No